CLINICAL TRIAL: NCT02638012
Title: Prospective Pilot Study of Floseal for the Treatment of Anterior Epistaxis in Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Prospective Pilot Study of Floseal for the Treatment of Anterior Epistaxis in Patients With (HHT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-057
Record Dates: First submitted 2015-10-13; First posted 2015-12-22 (Estimated); Results first posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT); Epistaxis
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — FloSeal Matrix; Drug Packaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HHT - Floseal (Experimental): Once the bleeding has stopped following application of the Floseal® a 50 cc syringe with sterile saline will be used to irrigate the treated nasal cavity to remove any excess Floseal® product as per manufacturer recommendations. This is done with the patient's head tilted downwards at a 30 degree angle so that the irrigation and excess product is removed from the nasal cavity.
  If bleeding is not controlled after up to two Floseal applications, the gel and clots will be removed with suction, and the patient will be treated with a standard packing treatment (standard of care).
  Interventions: Drug: Floseal; Other: Packing

INTERVENTIONS:
Drug: Floseal — Topical lidocaine spray (2%) is then administered using 1-2 sprays in the affected nasal cavity via the nostril that is to have Floseal® applied. Once the bleeding has stopped following application of the Floseal® a 50 cc syringe with sterile saline will be used to irrigate the treated nasal cavity to remove any excess Floseal® product as per manufacturer recommendations. This is done with the patient's head tilted downwards at a 30 degree angle so that the irrigation and excess product is removed from the nasal cavity. Once the irrigation is complete, the nasal cavity is inspected for evidence of continued bleeding.
  Other Names: Floseal hemostatic matrix
Other: Packing — If bleeding is not controlled after up to two Floseal applications, the gel and clots will be removed with suction, and the patient will be treated with a standard packing treatment (standard of care).

SUMMARY:
Current management strategies for severe and recurrent epistaxis secondary to Hereditary hemorrhagic telangiectasia (HHT) include surgical procedures, and uncomfortable nasal packing, both of which are often only short-term solutions. Floseal® may provide a non-invasive and less painful treatment option for epistaxis in HHT patients. This hemostatic agent has been shown to be an effective intraoperative hemostatic agent in a number of surgical procedures including endoscopic sinus surgery. It has also been shown to be favorable over nasal packing at controlling acute anterior epistaxis. Though the efficacy of using Floseal® for epistaxis in HHT patients has been proven anecdotally in the literature it has yet to be proven in a prospective clinical trial. The results of this pilot study will provide insight into the efficacy of using Floseal® in the management of severe epistaxis in HHT patients and to assist in the development of a full-scale prospective clinical trial.

DETAILED DESCRIPTION:
Hereditary hemorrhagic telangiectasia (HHT), also known as Osler-Weber-Rendu syndrome, is an autosomal dominant disorder that is characterized by abnormal blood vessel development. This dysplasia manifests as mucocutaneous telangiectases and visceral arteriovenous malformations (AVM).

The most common symptom is epistaxis occurring secondary to telangiectases in the nasal mucosa in more than 90% of HHT patients. Heterogeneity exists in the severity of epistaxis experienced by HHT patients; therefore, treatments and management strategies can vary. For minor bleeding, conservative management may include preventing drying of the nasal mucosa with the use of ointments and humidification. In some cases, topical or systemic estrogen may also be used to improve the stability of the nasal mucosa, thereby reducing bleeding. Commonly, anterior nasal packing is used as a non-surgical management strategy to control major bleeding. When medical management strategies have failed, laser coagulation of the telangiectases or septodermoplasty may be considered however, these solutions are temporary as telangiectasia are known to recur. In the acute setting, embolization may be used to occlude the abnormal vasculature while maintaining blood flow to the surrounding tissue; however, this is also not an effective long-term solution. Severe and difficult to manage epistaxis has been effectively treated using the modified Young's procedure where closure of the nostril is achieved by suturing together circumferential skin and mucosa flaps.

Floseal hemostatic matrix (Floseal®) is a hemostatic agent that consists of two major components. The first are gelatin granules that swell when they come into contact with blood or other wet surfaces creating a tamponade effect. The second is a high concentration of human thrombin that promotes natural clot formation by converting fibrinogen to fibrin. Floseal® is hydrophilic and therefore adheres well to wet tissues. It is indicated for use as an adjunct surgical hemostat and it has recently been demonstrated to be an effective treatment for epistaxis. A prospective, randomized, controlled trial compared Floseal® to nasal packing in the treatment of acute anterior epistaxis. The results showed Floseal® to be better at initially controlling epistaxis and resulted in fewer rebleed events within a seven day follow-up period. Patients also reported less pain and greater overall satisfaction with Floseal® as compared with nasal packing. Similarly, two prospective studies have evaluated the use of Floseal® for the treatment of posterior epistaxis. These trials also showed Floseal® treatment to be an effective treatment for posterior epistaxis. Furthermore, the use of Floseal® was associated with substantial institutional cost savings.

In summary, Floseal® has been demonstrated to be an effective treatment for posterior epistaxis, regardless of origin within the nose. Recently, Floseal® has been used in patients with HHT. This case series showed that patients with anterior epistaxis due to HHT could self-administer Floseal® to treat recurrent anterior epistaxis at their home without a contact with the medical system, as would customarily occur. This directly leads to an improvement in the quality of life of the patients in this study. Impairment of the quality of life for patients with HHT is a significant concern. Compared to the normative population, all subscales of SF36, but bodily pain, have been shown to be significantly poorer in the HHT patients. Studies of HHT substantiate that disease severity is associated with poorer QoL in these patients. Treatments for epistaxis that can improve the quality of life for patients with HHT are needed.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of HHT
* Active anterior epistaxis

Exclusion Criteria:

* A known sensitivity to any of the materials of Floseal® or the topical medications administered as part of the evaluation and treatment of epistaxis (lidocaine, xylometazoline hydrochloride)
* Pregnant and/or breast feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12; Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lee, MD, MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharathkumar AA, Shapiro A. Hereditary haemorrhagic telangiectasia. Haemophilia. 2008 Nov;14(6):1269-80. doi: 10.1111/j.1365-2516.2008.01774.x. PMID 19141168
- [Background] Olitsky SE. Hereditary hemorrhagic telangiectasia: diagnosis and management. Am Fam Physician. 2010 Oct 1;82(7):785-90. PMID 20879701
- [Background] Pau H, Carney AS, Murty GE. Hereditary haemorrhagic telangiectasia (Osler-Weber-Rendu syndrome): otorhinolaryngological manifestations. Clin Otolaryngol Allied Sci. 2001 Apr;26(2):93-8. doi: 10.1046/j.1365-2273.2001.00442.x. PMID 11309047
- [Background] Mathiasen RA, Cruz RM. Prospective, randomized, controlled clinical trial of a novel matrix hemostatic sealant in patients with acute anterior epistaxis. Laryngoscope. 2005 May;115(5):899-902. doi: 10.1097/01.MLG.0000160528.50017.3C. PMID 15867662
- [Background] Hoag JB, Terry P, Mitchell S, Reh D, Merlo CA. An epistaxis severity score for hereditary hemorrhagic telangiectasia. Laryngoscope. 2010 Apr;120(4):838-43. doi: 10.1002/lary.20818. PMID 20087969
- [Background] Kilty SJ, Al-Hajry M, Al-Mutairi D, Bonaparte JP, Duval M, Hwang E, Tse D. Prospective clinical trial of gelatin-thrombin matrix as first line treatment of posterior epistaxis. Laryngoscope. 2014 Jan;124(1):38-42. doi: 10.1002/lary.24240. Epub 2013 Jun 28. PMID 23754469
- [Background] Warner L, Halliday J, James K, de Carpentier J. Domiciliary floseal prevents admission for epistaxis in hereditary hemorrhagic telangiectasia. Laryngoscope. 2014 Oct;124(10):2238-40. doi: 10.1002/lary.24701. Epub 2014 May 2. No abstract available. PMID 24706356
- [Background] Geirdal AO, Dheyauldeen S, Bachmann-Harildstad G, Heimdal K. Quality of life in patients with hereditary hemorrhagic telangiectasia in Norway: a population based study. Am J Med Genet A. 2012 Jun;158A(6):1269-78. doi: 10.1002/ajmg.a.35309. Epub 2012 Apr 23. PMID 22529055
- [Background] Geisthoff UW, Heckmann K, D'Amelio R, Grunewald S, Knobber D, Falkai P, Konig J. Health-related quality of life in hereditary hemorrhagic telangiectasia. Otolaryngol Head Neck Surg. 2007 May;136(5):726-33; discussion 734-5. doi: 10.1016/j.otohns.2006.12.019. PMID 17478205
- [Background] Jameson M, Gross CW, Kountakis SE. FloSeal use in endoscopic sinus surgery: effect on postoperative bleeding and synechiae formation. Am J Otolaryngol. 2006 Mar-Apr;27(2):86-90. doi: 10.1016/j.amjoto.2005.07.011. PMID 16500469
- [Derived] Lee JM, Wu V, Faughnan ME, Lasso A, Figol A, Kilty SJ. Prospective pilot study of Floseal(R) for the treatment of anterior epistaxis in patients with hereditary hemorrhagic telangiectasia (HHT). J Otolaryngol Head Neck Surg. 2019 Oct 15;48(1):48. doi: 10.1186/s40463-019-0379-y. PMID 31615556

RESULTS

PARTICIPANT FLOW:
Groups:
- Floseal Treatment: All patients within the Floseal treatment group received a total of 5 mL of Floseal (one standard preparation), applied under direct visualization into the affected nasal cavity using the provided application catheter.
Period: Overall Study
Arm/Group | Floseal Treatment
Started | 8
Completed | 7
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Floseal Treatment: Patient baseline characteristics
Arm/Group | Floseal Treatment
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 7

OUTCOME MEASURES:

1. Primary Outcome: Epistaxis Severity Score (ESS)
Description: Questions include:
  1. How often did you typically have nosebleeds during the past one month?
  2. How long did each nosebleed typically last for you during the past one month?
  3. How would you describe your typical nosebleed intensity during the past one month?
  4. Have you sought medical attention outside of this research study for your nosebleeds during the past one month?
  5. Are you anemic currently?
  6. Have you received a red blood cell transfusion specifically for nosebleeds during the past month?
  The responses to each of the six questions are assigned a weighted integer that is multiplied by the question's coefficient. These are added to yield the raw score, which is then normalized by dividing by the maximum possible score, then multiplied by 10 to give the normalized score. Range of normalized score is 0 to 10. With 0 representing low severity, and 10 representing high severity.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Floseal Treatment
Number analyzed (Participants) | 7
score on a scale
  Baseline | 5.13 (3)
  1 month follow up | 3 (3.13)

2. Secondary Outcome: Change in Number of Nose Bleeds During One Month Period Following Treatment
Time Frame: Baseline and 1 month
Population: Data was incomplete or unavailable for all participants and so this outcome measure was not recorded.
Arm/Group | Floseal Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Severity Rating of Nose Bleeds During One Month Period Following Treatment
Description: Questionnaire asks: 1) date, 2) number of nosebleeds, 3) average nosebleed severity (scale of 0 to 10, 10 being as worse as it can be)
Time Frame: Baseline and 1 month
Population: Data was incomplete or unavailable for all participants and so this outcome measure was not recorded.
Arm/Group | Floseal Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Need for Additional Interventions to Control Epistaxis During One Month Following Floseal® Application
Time Frame: Baseline and 1 month
Population: Data was incomplete or unavailable for all participants and so this outcome measure was not recorded.
Arm/Group | Floseal Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Clinical Assessment of Telangiectases, Crusting, Scarring, and Active Bleeding Sites in the Nasal Cavity Before and One Month Following Treatment
Description: Clinical assessment score of 1) nasal telangiectases, 2) crusting, 3) scarring, and 4) active bleeding sites. Each side of the nose is scored independently from 0 - none to 10 - severe. Range of the total score is from 0 to 80.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Floseal Treatment
Number analyzed (Participants) | 7
score on a scale
  Baseline | 17.29 (7.70)
  1 month follow up | 9.57 (7.81)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Floseal Treatment
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT02638012/Prot_SAP_000.pdf